CLINICAL TRIAL: NCT03700151
Title: Efficacy of an Intervention for the Children With Severe Speech Sounds Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Michael Tong, Chairman, Department of Otorhinolaryngology, Head and Neck Surgery, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPF18HLF26
Record Dates: First submitted 2018-09-22; First posted 2018-10-09 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Speech Sound Disorder; Apraxia of Speech; Developmental Verbal Dyspraxia
MeSH Terms: conditions — Speech Sound Disorder; Apraxias | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A group of 20 participants with severe speech sound disorders will receive the proposed intervention. Pre- and post-test data will be collected to study the treatment efficacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with SSD (Experimental): Participants will receive a piloted treatment programme for children with severe speech sound disorders, especially childhood apraxia of speech.
  Interventions: Behavioral: Treatment for Children with Severe Speech Sound Disorders

INTERVENTIONS:
Behavioral: Treatment for Children with Severe Speech Sound Disorders — The intervention has two tasks, including syllable repetition tasks which requires participants to repeat nonsense syllables, and training of vocabulary or phrase with the application of Principle of Motor Learning.

SUMMARY:
Speech sound disorders (SSDs) is one type of communication problems in children. It is a board term describing different difficulties that impact speech intelligibility. There are different types of SSDs, including motor-based disorders (e.g., dysarthria and childhood apraxia of speech [CAS]), structurally based disorders (e.g., cleft-palate), syndrome/condition-related disorders (e.g., Down), sensory-based conditions (e.g., hearing loss), and idiopathic in nature.

Among different types of SSDs in children, childhood apraxia of speech (CAS) is a type of motor speech disorders with symptom complex, and is always considered as severe SSDs if objective measurement of severity, percentage of consonant correct (PCC) is applied.

Evidence of different intervention approaches of CAS and SSDs have been obtained from English-speaking children. This is unknown if these approaches can be applied to languages which are different from English in terms of the sound inventory and prosody.

A treatment program for Cantonese-speaking children with childhood apraxia of speech was studied. Preliminary positive findings were obtained from two participants in an ABA single-case study. With the preliminary positive data, a higher level of evidence could be obtained from group study. The purpose of this study is to determine the efficacy of the proposed intervention for children with severe SSDs by quasi-experimental design.

DETAILED DESCRIPTION:
A treatment program for children with severe SSDs, especially childhood apraxia of speech (CAS), a type of motor speech disorders in children was proposed. The program includes syllable repetition tasks and training of core vocabularies. In the syllable repetition tasks, children are required to repeat nonsense syllables three to five times according to their sequencing abilities. This flexibility training of syllables was believed to address the underlying speech motor deficits of children with severe SSDs. The level of difficulty is increased in a systematic way to help progression of children speech skills. In the training of core vocabulary, ten vocabularies which have high functional values in children's daily communication were proposed by parents. Speech therapists are instructed to prioritize the vocabularies and practice the children with the application of Principle of Motor Learning (PML) and Dynamic Temporal and Tactile Cueing (DTTC).

Preliminary positive findings were obtained from two participants in an single-case study. The results showed that the treatment program was able to increase the number of syllable per words, increase the speech sound accuracy, increase the complexity of syllable structure, and increase speech intelligibility.

A quasi-experimental one-group pre- and post-test design will be conducted to study the efficacy of the proposed treatment. A power calculation has been used to determine the number of participants to be recruited. Preliminary findings of the proposed treatment program was obtained. One of the two participants demonstrated statistically significant differences with medium effect size. Based on this, with the estimated medium effect size (d =0.6) with .05 alpha error probability and 0.8 power (1-beta error probability), a total of 19 participants are required.

Twenty children aged between 3 to 18 will be recruited. The specific inclusion criteria of the participants are set as follow:

1. Cantonese as the main language input
2. No oral structural abnormality
3. No hearing loss
4. No diagnosis of Autism Spectrum Disorders
5. No major behavioral problem

Pre-treatment assessment and baseline probes:

Pre-treatment assessment will be implemented to all participants. The assessment protocol proposed by Wong (2017) will be used. The assessment protocol consists of case history taking, collecting speech sample, standardized language assessment, standardized speech screening, non-standardized motor speech assessment, hearing screening, tone identification test, and observation of suprasegmental features.

A specially designed word list will be used to take the baseline data for all children about their number of syllable in words, speech sound accuracy, complexity of phonotactic structure. Speech intelligibility will be measured by percentage of consonant correct (PCC) in the children's 15-minutes speech sample.

CAS diagnosis:

After the assessment, the speech therapists will make a diagnosis of CAS if applicable and plan the treatment goals for the children. The speech therapists will make a CAS diagnosis if the children show all 29 diagnostic clinical features of CAS proposed by Wong (2017). For planning treatment, the speech therapists will select stimuli for the syllable repetition task and discuss the core vocabularies with the parents for training.

Intervention:

Each participant will be allocated one or two trained speech therapists for all treatment sessions. All participants will receive the 45-minute sessions, twice a week for six weeks for a total of 12 treatment sessions. All the sessions will be video-recorded for measurement of treatment fidelity. The detail of the treatment protocol was documented in Wong (2017).

In-session probes:

Speech therapists will require the children to produce the word lists at the end of every six sessions of treatment. Two probe sessions will be taken after the practice at 6th and 12th session.

Post-treatment evaluation:

All children will be required to produce the specially designed words lists and be collected a 15-minute speech sample by speech therapists one week after the end of 12th treatment session to document the post-treatment performances in term of the number of syllable in words, speech sound accuracy, phonotactic complexity and speech intelligibility.

Data Analysis:

The pre- and post-treatment differences of the percent correct of the speech sound accuracy and speech intelligibility will be compared by the Wilcoxon Signed-Rank Test. It is hypothesized that the treatment group will show significant improvement on the two outcome measures after intervention.

The inter-rater and intra-rater reliability of the judgement on CAS diagnosis will be analysed by Cohen's kappa. The assessor and the video-viewer will re-view 20% of the videos that were viewed for CAS diagnosis one month later to determine the intra-rater reliability. Another 20% of the rated data will be randomly selected to compare and determine the inter-rater reliability.

A training workshop will be given to the speech therapists who will provide intervention for the children prior to the start of intervention. A checklist will be used to measure the fidelity of the intervention. The measures consist of 1) application of the program structure, including, timing, sequences and content of the tasks, and 2) application of the cueing hierarchy, provision of feedback and the proposed practice amount. Two independent speech therapists will randomly view 20% of all treatment sessions and rate the fidelity by the checklist. The intra-rater and inter-rater reliability of the rating will be measured by Cohen's kappa.

ELIGIBILITY:
Inclusion Criteria:

- Aged between 3 to 18 Cantonese as the main language input No oral structural abnormality No hearing loss No diagnosis of Autism Spectrum Disorders No major behavioural problem

Exclusion Criteria:

-

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Percent correct for target speech sounds | 6 weeks treatment

SECONDARY OUTCOMES:
Speech intelligibility | 6 weeks treatment
  5-point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No